CLINICAL TRIAL: NCT06278727
Title: Development and Validation of the Prediction Model for Functional Mitral Regurgitation Regression in Heart Failure Patients Taking Guideline-directed Medical Therapy
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1173-01
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mitral Regurgitation; Heart Failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors; Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regression group: Regression group contains the patients whose FMR regresses after taking GDMT for at least 3 months.
  Interventions: Drug: angiotensin-converting enzyme inhibitors/angiotensin II receptor blocker/angiotensin receptor-neprilysin inhibitor; Other: The development of the prediction model
- No-reaction group: No-reaction group contains the patients whose FMR has no regression by every clinical visit.
  Interventions: Drug: angiotensin-converting enzyme inhibitors/angiotensin II receptor blocker/angiotensin receptor-neprilysin inhibitor

INTERVENTIONS:
Drug: angiotensin-converting enzyme inhibitors/angiotensin II receptor blocker/angiotensin receptor-neprilysin inhibitor — Guideline-directed Medical Therapy (GDMT) includes those 4 drugs, and only taking at least 3 drugs could be recognized as GDMT.
  Other Names: beta-blockers; mineralcorticoid recept antagonist; sodium-glucose linked transporter-2 inhibitor
Other: The development of the prediction model — The prediction model of FMR regression would be developed to recognize patients whose FMR would regress due to GDMT, and consequently help determine the treatment.
  Groups: Regression group

SUMMARY:
This observational study is to develop and validate the prediction model for functional mitral regurgitation regression in heart failure patients taking GDMT. The patients diagnosed ≥2+ functional mitral regurgitation by ultrasonic cardiogram are enrolled in this study and would be clinically followed by at least one year (clinical visit at 3 months, 6 months, and 12 months), and then by when the endpoints are reached.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* ≥2+ FMR
* Receiving GDMT

Exclusion Criteria:

* degenerative mitral regurgitation
* myocardial infarction, percutaneous coronary intervention, coronary bypass grafting surgery, cardiac resynchronization therapy, or stroke within three months prior to this study
* ≥2+ aortic stenosis or regurgitation
* previous surgical mitral valve repair or replacement
* restrictive cardiomyopthy, hypertrophic cardiomyopathy, or constrictive pericarditis
* severe heart failure (NYHA class IV) or left ventricular ejection fraction < 20%
* symptomatic hypotension affecting GDMT prescription
* severe hepatic or renal insufficiency
* life expectancy < 12 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FMR regression rate | 3 months
  the rate of FMR regression by at least 1 grade by 3 months

SECONDARY OUTCOMES:
FMR regression rate | 6 months
  the rate of FMR regression by at least 1 grade by 6 months
composite endpoint | one year
  the composite endpoint includes all-cause mortality, worsening heart failure, and mitral intervention. The worsening heart failure includes heart failure hospitalization, NYHA cardiac function upgrades ≥1 grade, and acute heart failure needing diuretic or outpatient adjustment of prescription.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun-Yatsen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided